CLINICAL TRIAL: NCT01679574
Title: Letrozole Versus Clomiphene Citrate Plus Metformin in the First Treatment of Infertility in Patients With Polycystic Ovarian Syndrome
Brief Title: Letrozole or Combined Clomiphene Citrate Metformin as a First Line Treatment in Women With Polycystic Ovarian Syndrome
Acronym: PCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, ahmed ali, Prinicple investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pcolcm
Record Dates: First submitted 2012-08-31; First posted 2012-09-06 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCO
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Letrozole; Clomiphene; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- letrozole (Experimental): Letrozole tablets (Femara; Novartis Pharma, Switzerland) 2.5 mg letrozole daily from day 3 of the menses for 5 days
  Interventions: Drug: Letrozole
- Metformin and clomiphene (Active Comparator): .Drug: metformin (Cidophage®; CID,Cairo, Egypt) metformin 1500 daily for 3 months
  * Drug: CC (Clomid®; Global Napi Pharmaceuticals, Cairo, Egypt) 100 mg CC for 5 days starting from day 3 of menstruation
  Interventions: Drug: Clomiphene; Drug: Metformin

INTERVENTIONS:
Drug: Letrozole — •Drug: Letrozole tablets (Femara; Novartis Pharma, Switzerland) 2.5 mg letrozole daily from day 3 of the menses for 5 days
  Other Names: Femara; Novartis Pharma, Switzerland
  Arms: letrozole
Drug: Clomiphene — •Drug: CC (Clomid®; Global Napi Pharmaceuticals, Cairo, Egypt) 100 mg CC for 5 days starting from day 3 of menstruation
  Other Names: clomid
  Arms: Metformin and clomiphene
Drug: Metformin — •Drug: metformin HCl (Cidophage®; CID,Cairo, Egypt) metformin HCl 1500 daily for 3 months
  Other Names: Cidophage
  Arms: Metformin and clomiphene

SUMMARY:
The purpose of this study is to compare and determine the efficacy of letrozole administration to that of combined metformin and Clomiphene in infertile women with polycystic ovary syndrome (PCOS) not treated before with any ovulation induction agent

DETAILED DESCRIPTION:
The study will be in 200 patient diagnosed to have PCOS among those attending the Fertility Outpatient Clinic at the Women's Health Center, Assiut University Hospitals.

The present study was prospective randomized controlled trial conducted over a period of 3 years from 1st of January 2009 to 1st of January 2012, at the Women's Health Center, Assiut University hospital, Assiut, Egypt, after approval was received from the Ethics Committee of faculty of medicine , Assiut University. Women referred to the infertility clinic in women's health center were screened for PCO using Rotterdam consensus criteria for the diagnosis of PCOS. The patients who were newly diagnosed as PCO and not treated previously were invited to participate in our study. Written informed consent was obtained from each participant after an information sheet had been provided. The patients had the right to refuse participation in the study or to withdraw at any time without being denied their full regular clinical care. All personal information and medical data were confidential and were not made available to third parties. All participants met the Rotterdam consensus criteria for the diagnosis of PCOS. At admission, a thorough medical history was taken and all women underwent physical examination, which included anthropometric measurements and after spontaneous menstruation or progestin induced withdrawal bleeding, basal endocrine evaluation on day 3 of the cycle included measurement of the serum concentrations of luteinizing hormone (LH), follicle-stimulating hormone (FSH),thyroid stimulating hormone(TSH ) and prolactin. Then vaginal sonographic examination were done to measure endometrial thickness and exclude cases endometrial pathology or baseline ovarian cysts.

The participants were randomized to receive letrozole or clomiphene citrate plus metformin. Randomization was performed using a computer-generated random numbers table, and allocation concealment was achieved using serially numbered opaque envelopes that were only opened once the interventions were assigned.

In the letrozole group, the ovaries were stimulated using 2.5mg/day letrozole (Femara; Novartis Pharma, Basel, Switzerland) for 5 days,in the form of one tablet( 2.5 mg) per day for 5 days from day 3 to day 7 of the menstrual cycle and if ovulation has occurred with no pregnancy continue on the same dose for another 2 consecutive cycles ,but if no ovulation increase the dose to 2 tablets per day(5 mg) for another 2 consecutive cycles in the same manner .

The patients in the second group will take metformin (Cidophage tablets,500 mg per tablet; CID, ARE, in an oral dose of 1,500 mg/d) 500mg three times daily for 3 months Plus clomid(50-mg tablets twice daily; Global Napi Pharmaceuticals, Cairo, Egypt , Arab Republic of Egypt) In the form of 50 mg twice daily (100mg /day) for 5 days from day 3 to day 7 of menstrual cycle and to be repeated for 3 consecutive cycles in the same manner if no pregnancy occur.

In both groups, endometrial thickness and mean follicular diameter were assessed by the same investigator using transvaginal ultrasound on days 2 ,10, 12, and 14 of the menstrual cycle, and 10 000 IU of human chorionic gonadotropin (hCG) (Pregnyl; Organon, Oss, The Netherlands) were injected intramuscularly if there was at least 1 leading follicle measuring 18 mm or more in diameter and endometrial thickness detected at that time(endometrial thickness was determined at the greatest diameter perpendicular to the midsagittal plane in the fundal region, including both layers of the endometrium). All participants were advised to have intercourse 24-36 hours after the hCG injection. Two days after being given Human chorionic gonadotropin, the patients were assessed for signs of ovulation (disappearance of preovulatory follicle, fluid in the cul-de-sac, and/or corpus luteum formation). Pregnancy will be diagnosed when positive pregnancy test in urine done or a gestational sac was detected on transvaginal ultrasound examination 1week after the missed period or serum β-hCG concentration 14 days after HCG injection if menses had not occurred. A biochemical pregnancy was considered when the serum β-hCG concentration was 50 mIU/mL or more in the absence of menstruation. All study medication were stopped when there was positive pregnancy test.Pregnant patients then will be followed up until an ultrasound could document the viability of pregnancy. A clinical pregnancy was defined as the presence of a gestational sac with a beating fetal heart on transvaginal ultrasound. A spontaneous abortion was defined as the spontaneous loss of a pregnancy before the end of the 20th week.

ELIGIBILITY:
Inclusion Criteria:

* All participants met the Rotterdam consensus criteria for the diagnosis of PCOS . .Primary infertility because of anovulation for at least 1 year.
* Only fresh (not treated previously) cases were recruited. .The male partner of each participant was required to have a normal result on semen analysis (count>20million/ml,motility>40%and normal morphology >30%).
* Each woman was required to have patent tubes on hysterosalpingography or on a diagnostic laparoscopy.

Exclusion Criteria:

* Age below 18 years or above 35 years , trial of ovulation induction prior to the stud ,BMI >35 .
* Presence of other causes of infertility; hyperprolactinemia (morning plasma prolactin concentration 30 ng/mL or more); any other endocrine, hepatic, or renal disorder; presence of an organic pelvic mass;
* History of abdominal surgery that might have caused pelvic factor infertility.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2009-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
ovulation rate | 3 years
  Principally the ovulation rate as well as the number of growing and mature follicles and endometrial thickness (mm).

SECONDARY OUTCOMES:
The occurrence of pregnancy and miscarriage | 3 years
  The occurrence of pregnancy and miscarriage

CONTACTS AND LOCATIONS:
Overall Officials: Tarek al Hussaini, prof, Study Chair — Assiut University; Safowt Abd El Rady, Prof, Study Director — Assiut university hosiptal; Mohamad S Abd Allah, Ass prof, Study Director — assiut university hosital
Locations (1):
- Assiut University, Asyut, Asyut Governorate, Egypt